CLINICAL TRIAL: NCT01741987
Title: An Effectiveness of Osmoprotective Containing Lubricants in Dysfunctional Tear Syndrome (DTS) and Post Refractive Surgery Patients
Brief Title: Osmoprotective Containing Lubricants in Dysfunctional Tear Syndrome and Post Refractive Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rossen Mihaylov Hazarbassanov, MD, PhD, MD, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1346/08
Record Dates: First submitted 2012-11-27; First posted 2012-12-05 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Dry Eye; Ametropia
MeSH Terms: conditions — Dry Eye Syndromes; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- optive® eye drop (Active Comparator)
  Interventions: Other: Fresh Tears ®
- fresh tears ® eye drop (Placebo Comparator)
  Interventions: Other: Optive ®

INTERVENTIONS:
Other: Optive ® — instilation of 1 drop each eye 4 times per day
  Arms: fresh tears ® eye drop
Other: Fresh Tears ® — instilation of eye drop 4 times a day (qid)
  Arms: optive® eye drop

SUMMARY:
The purpose of this project is to determine the effectiveness of an eyewash osmoprotective lubricant comparing to castor oil containing and non-osmoprotective lubricants in different types of DTS and post refractive surgery patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients willing and able to comply with the protocol who are not planning changes in diet, topical or systemic drugs during the course of study.
2. DTS all the patients will be diagnosed for mild to moderate evaporative dry eye as defined by following criteria that will be given by Outcome measurements:

   2.1. Break up time. 2.2. Lissamine green staining. 2.3. OSDI and Patient Symptomatology Questionnaire.
3. The patients, whose are going to be submitted for refractive surgery.

Exclusion Criteria:

1. Any patient with punctual occlusion or punctual plugs.
2. Patients with active ocular infection or inflammatory disease, history of herpetic keratitis, history of retinal detachment, concurrent contact lens use during trial period,
3. Patients with glaucoma, anterior membrane dystrophy, active trichiasis or any eyelid globe malposition abnormality.
4. Patients with Epiphora.
5. Patients must not have participated in any investigational therapeutic drug or device trial within the 30 days prior to their start date for this trial.
6. Any patient suffering from organic brain syndromes or major psychiatric disorder that would interfere with compliance or subjective reporting will be discouraged from participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
patients satisfaction with osmoprotective lubricant on different types DTS. | 3 months

SECONDARY OUTCOMES:
Our purpose is to determine the differential effects of Optive® castor oil Endura ® on different types DTS. | 3 months
Physician satisfaction with Optive® | 3 months

OTHER OUTCOMES:
Our purpose is to determine the differential effects of Optive® vs. FreshTears ® on post refractive surgery patients. | 3 monthas
change from baseline in Ocular Surface Disease Index (OSDI) | 3 moths
change from baseline in tear break up time (BUT) | 3 mothas
change from baseline in lissamine green staining | 3 months
change form baseline in impression cytology | 3 months
change from baseline in tear osmolarity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rossen M Hazarbassanov, MD, Principal Investigator — Department of Ophtahlmology, UNIFESP& EPM, Sao Paulo, SP, Brazil
Locations (1):
- Department of Ophthalmology, UNIFESP&EPM, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: eye diseases — http://www.nlm.nih.gov/medlineplus/eyediseases.html
- See also: FDA Resources on Drugs and Devices — http://clinicaltrials.gov/ct2/info/fdalinks